CLINICAL TRIAL: NCT03288038
Title: A Multi-center, Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy of Rosuvastatin and Ezetimibe and Rosuvastatin Monotherapy in Patients With Primary Hypercholesterolemia
Brief Title: The Efficacy and Safety of Combination Therapy of Rosuvastatin and Ezetimibe and Rosuvastatin Monotherapy in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SP-RE-003
Record Dates: First submitted 2017-08-18; First posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RSV5mg + EZE 10mg (Experimental): Rosuvastatin 5mg/Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- RSV5mg (Active Comparator): Rosuvastatin 5mg
  Interventions: Drug: Rosuvastatin
- RSV10mg + EZE10mg (Experimental): Rosuvastatin 10mg/ Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- RSV10mg (Active Comparator): Rosuvastatin 10mg
  Interventions: Drug: Rosuvastatin
- RSV20mg + EZE10mg (Experimental): Rosuvastatin 20mg/Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- RSV20mg (Active Comparator): Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin
Drug: Ezetimibe
  Arms: RSV10mg + EZE10mg; RSV20mg + EZE10mg; RSV5mg + EZE 10mg

SUMMARY:
A Multi-center, Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy of Rosuvastatin and Ezetimibe and Rosuvastatin Monotherapy in Patients with Primary Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Patients with primary hypercholesterolemia
3. Patients who were informed about the purpose, method, effects, risks of this clinical study and have provided a written consent form signed by him/herself or by a representative
4. those who show an LDL-C level of 250 mg/dL or below and a TG level of less than 350 mg/dL at the run-in period (Week -1), and fall under the criterion of requiring the administration of antidyslipidemic drug of NCEP ATP III

Exclusion Criteria:

1. Patients with hypersensitivity to the investigational product or its ingredients
2. Those with an uncontrolled hypertension (SBP ≧ 180 mmHg or DBP ≧ 100 mmHg)
3. Those with a history of unstable angina, myocardial infarction, transient ischemic attack, cerebral vascular disease, coronary artery bypass or coronary intervention within 3 months of screening date
4. Those with a history of malignant tumor within 5 years
5. Those with a history of myopathy or rhabdomyolysis
6. Those who show clinically significant confirmed laboratory test results (1) Patients showing AST or ALT level of greater than 2 times the institutional upper limit of normal or those with active liver disease or chronic hepatitis (2) A serum creatinine level greater than 2 times the institutional upper limit of normal (3) HbA1c > 9% (4) Those with TSH level of greater than 1.5 times the institutional upper limit of normal (5) Those with CK level greater than 2 times the institutional upper limit of normal (However, except for an increase caused by a recent trauma, intramuscular injection or strenuous exercise)
7. Those who were given, within 4 weeks prior to the baseline (8 weeks in case of fibrate) or are expected to be given during the study period, a drug that can have an effect on the efficacy assessment of the clinical study (eg: antidyslipidemic drug (statins, ezetimibe, fibrates, BAS, nicotinic acid and derivative, etc.), systemic glucocorticosteroids, steatolytic enzyme inhibitor, cyclosporine, HIV proteinase inhibitor, macrolide class antibiotics, etc.)
8. Patients who were given estrogen within 3 months from the screening or those who are expected to be given an administration during the study period. (However, a patient who is under a hormone replacement therapy (HRT) will be allowed if no dose change is expected in the course of the clinical study.)
9. Those with a history of alcohol or drug abuse
10. Patients with a hereditary disorder of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
11. Pregnant or breast-feeding women
12. Women of childbearing potential or men who do not intend to use an adequate contraceptive measure during the study period and for 4 weeks after the end of the study(Adequate contraception: Administration and transplantation of a progestin-only contraceptive pill, intrauterine device, condom, spermicidal agent, etc.)
13. Patients who participated in another clinical study within 3 months from the screening date or have not had a washout period of at least 5 times the half-life of the active ingredient of the previously administered investigational product, whichever is longer
14. Those with drug malabsorption
15. Patients who has been judged by the investigator to be ineligible to participate in the clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 8 week in LDL-Cholesterol | baseline and 8 week

SECONDARY OUTCOMES:
Percent change from baseline to 4 week in LDL-Cholesterol | baseline and 4 week
The change in the LDL-C level from the baseline to Week 4 and Week 8 | baseline to 4 and 8 week
The change and percent change in the levels of TC, TG, HDL-C, non-HDL-C, apolipoprotein B, and hs-CRP from the baseline to Week 4 and Week 8 | baseline to 4 and 8 week
The change and percent change in the ratios of LDL-C/HDL-C, TC/HDL-C, non-HDL-C/HDL-C, and Apo B/Apo A-I from the baseline to Week 4 and Week 8 | baseline to 4 and 8 week
The ratio of the subjects who have reached the target LDL-C level according to the NCEP ATP(National Cholesterol Education Program Adult Treatment Panel) III Guideline at Week 4 and Week 8 | baseline to 4 and 8 week

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Dongguk University Ilsan Hospital, Goyang-si
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Boramae Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - KyungHee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim W, Yoon YE, Shin SH, Bae JW, Hong BK, Hong SJ, Sung KC, Han SH, Kim W, Rhee MY, Kim SH, Lee SE, Hyon MS, Hwang GS, Son JW, Kim JY, Kim MK, Kim SW, Park JH, Shin JH, Park CG. Efficacy and Safety of Ezetimibe and Rosuvastatin Combination Therapy Versus Those of Rosuvastatin Monotherapy in Patients With Primary Hypercholesterolemia. Clin Ther. 2018 Jun;40(6):993-1013. doi: 10.1016/j.clinthera.2018.04.015. Epub 2018 May 30. PMID 29857919